CLINICAL TRIAL: NCT03546166
Title: Open, Prospective, Single-center Study Evaluating the Efficacy and Safety of 0.05% Ingenol Mebutate (Picato® 500) in the Treatment of Basal Cell Carcinoma
Brief Title: Study Evaluating the Efficacy and Safety of 0.05% Ingenol Mebutate (Picato® 500) in the Treatment of Basal Cell Carcinoma
Acronym: PICABAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-PP-21
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma
Keywords: basal cell carcinoma
MeSH Terms: conditions — Carcinoma; Carcinoma, Basal Cell | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TREATMENT (Experimental)
  Interventions: Drug: Picato 0.05% Topical Gel

INTERVENTIONS:
Drug: Picato 0.05% Topical Gel — apply on and 1 cm around the lesion, 0.47 g of Picato® gel 150 µg/g, once a day on 2 consecutive days. In case of treatment failure after 3 months, apply again on and 1 cm around the lesion, 0.47 g of Picato® gel 150 µg/g, once a day on 2 consecutive days.

SUMMARY:
Basal cell carcinomas (BCCs) are the most common form of cancer. The treatment of BCC can be surgical or topical for the low-risk subtypes. Topical treatments used for BCC are imiquimod and photodynamic therapy (PDT). Ingenol mebutate could provide a fast and easy topical therapy for BCC. Data regarding the treatment of BCC with ingenol mebutate are still limited. The investigators propose a pilot study to investigate the efficacy of 1 or 2 courses of ingenol mebutate 0,05%, on superficial and nodular BCC

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confi rmed, primary, previously untreated, nodular or superfi cial basal-cell carcinoma not arising on the face or scalp, measuring 1 to 4 cm (large axis)

Exclusion Criteria:

* Basal cell carcinomas of the scalp
* Basal cell carcinomas recurrent, sclerodermiform, infiltrant, metatypic
* Allergic patient to treatment products
* Patient treated with immunosuppressants, immunomodulators, systemic cytotoxic agents or local corticosteroids applied in the CBC area during the 4 weeks prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy, in terms of complete remission, of 1 of a topical treatment with picato 0.05% gel topical | 3 months
To evaluate the efficacy, in terms of complete remission, of 2 cycles (for patients who did not respond to the first cycle) of a topical treatment with picato 0.05% gel topical | 6 months

SECONDARY OUTCOMES:
determine the tolerance of the treatment: complete remission after 1 cycle | 3 months
  For patients in complete remission after 1 cycle
determine the tolerance of the treatment: complete remission after 2 cycle | 3 months and 6 months
  For patients in complete remission after 2 cycle
Evaluate the tumor response according to clinical criteria | 3 months
Evaluate the tumor response according dermoscopic, | 3 months
Evaluate the tumor response according Optical Coherence Tomography | 3 months
Evaluate the tumor response according ultrasound | 3 months
Evaluate the tumor response according histology | 3 months
Evaluate the tumor response according to clinical criteria | 6 months
  For patients in complete remission after 2 cycle
Evaluate the tumor response according to dermoscopic | 6 months
  For patients in complete remission after 2 cycle
Evaluate the tumor response according to Optical Coherence Tomography | 6 months
  For patients in complete remission after 2 cycle
Evaluate the tumor response according to ultrasound | 6 months
  For patients in complete remission after 2 cycle
Evaluate the tumor response according histology | 6 months
  For patients in complete remission after 2 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BAHADORAN, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsay JR, Suhrbier A, Aylward JH, Ogbourne S, Cozzi SJ, Poulsen MG, Baumann KC, Welburn P, Redlich GL, Parsons PG. The sap from Euphorbia peplus is effective against human nonmelanoma skin cancers. Br J Dermatol. 2011 Mar;164(3):633-6. doi: 10.1111/j.1365-2133.2010.10184.x. Epub 2011 Jan 27. PMID 21375515
- [Background] McKay KM, Sambrano BL, Fox PS, Bassett RL, Chon S, Prieto VG. Thickness of superficial basal cell carcinoma (sBCC) predicts imiquimod efficacy: a proposal for a thickness-based definition of sBCC. Br J Dermatol. 2013 Sep;169(3):549-54. doi: 10.1111/bjd.12402. PMID 23627639
- [Background] Mogensen M, Nurnberg BM, Forman JL, Thomsen JB, Thrane L, Jemec GB. In vivo thickness measurement of basal cell carcinoma and actinic keratosis with optical coherence tomography and 20-MHz ultrasound. Br J Dermatol. 2009 May;160(5):1026-33. doi: 10.1111/j.1365-2133.2008.09003.x. Epub 2009 Jan 12. PMID 19183171
- [Result] Prieto-Granada C, Rodriguez-Waitkus P. Basal cell carcinoma: Epidemiology, clinical and histologic features, and basic science overview. Curr Probl Cancer. 2015 Jul-Aug;39(4):198-205. doi: 10.1016/j.currproblcancer.2015.07.004. Epub 2015 Jul 8. No abstract available. PMID 26239203
- [Result] Williams HC, Bath-Hextall F, Ozolins M, Armstrong SJ, Colver GB, Perkins W, Miller PSJ; Surgery Versus Imiquimod for Nodular and Superficial Basal Cell Carcinoma (SINS) Study Group. Surgery Versus 5% Imiquimod for Nodular and Superficial Basal Cell Carcinoma: 5-Year Results of the SINS Randomized Controlled Trial. J Invest Dermatol. 2017 Mar;137(3):614-619. doi: 10.1016/j.jid.2016.10.019. Epub 2016 Dec 5. PMID 27932240
- [Result] Ogbourne SM, Suhrbier A, Jones B, Cozzi SJ, Boyle GM, Morris M, McAlpine D, Johns J, Scott TM, Sutherland KP, Gardner JM, Le TT, Lenarczyk A, Aylward JH, Parsons PG. Antitumor activity of 3-ingenyl angelate: plasma membrane and mitochondrial disruption and necrotic cell death. Cancer Res. 2004 Apr 15;64(8):2833-9. doi: 10.1158/0008-5472.can-03-2837. PMID 15087400
- [Result] Rosen RH, Gupta AK, Tyring SK. Dual mechanism of action of ingenol mebutate gel for topical treatment of actinic keratoses: rapid lesion necrosis followed by lesion-specific immune response. J Am Acad Dermatol. 2012 Mar;66(3):486-93. doi: 10.1016/j.jaad.2010.12.038. Epub 2011 Nov 4. PMID 22055282
- [Result] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- [Result] Siller G, Rosen R, Freeman M, Welburn P, Katsamas J, Ogbourne SM. PEP005 (ingenol mebutate) gel for the topical treatment of superficial basal cell carcinoma: results of a randomized phase IIa trial. Australas J Dermatol. 2010 May;51(2):99-105. doi: 10.1111/j.1440-0960.2010.00626.x. PMID 20546215